CLINICAL TRIAL: NCT01715207
Title: Comparison Study of the Effect of Aliskiren Versus Negative Controls on Aortic Stiffness in Patients With Marfan Syndrome Under Treatment With Atenolol
Brief Title: Comparison of Aliskiren vs Negative Controls on Aortic Stiffness in Patients With MFS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Duk-Kyung Kim, PhD, MD, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-10-025
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Marfan Syndrome
MeSH Terms: conditions — Marfan Syndrome | interventions — aliskiren; Atenolol

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atenolol & Aliskiren (Experimental): Atenolol tablet and Aliskiren 150mg or 300mg tablet by mouth per day for 6month
  Interventions: Drug: Aliskiren; Drug: Atenolol
- Atenolol (Other): Atenolol tablet(Negative controls, Open-label)
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Aliskiren
  Other Names: Rasilez
  Arms: Atenolol & Aliskiren
Drug: Atenolol
  Other Names: Tenormin

SUMMARY:
Marfan syndrome (MFS) is an inherited disorder of connective tissue with morbidity and mortality from aortic dilatation and dissection. The current standard of care is beta-blocker (BB) treatment and therapeutic target is heart rate. The degree of aortic dilatation and response to BB vary in adults with MFS. However, aortic stiffness is often present, and can be a predictor of aortic dilatation and cardiovascular complications. Aortic stiffness is a logical therapeutic target in adults with MFS.

Transforming growth factor beta(TGF-beta) mediates disease pathogenesis in MFS and contributes to aortic stiffness. Cross-talk between TGF-beta system and renin-angiotensin system (RAS) has been demonstrated. The angiotensin receptor blocker (ARB), losartan, inhibits TGF-beta activity and reverses aortic wall pathology in a Marfan mouse model. In a small cohort study, the use of ARB therapy (losartan or irbesartan) significantly slowed the rate of progressive aortic dilatation in patients with MFS, after BB therapy had failed to prevent aortic root dilatation. In another study, angiotensin converting enzyme inhibitor, perindopril, reduced both aortic stiffness and aortic root diameter in patients with MFS taking standard BB therapy. Renin inhibitor, aliskiren, has not been studied to reduce aortic stiffness and attenuate aortic dilatation in patients with MFS.

This trial is a randomized, open-label trial of 32 patients with Marfan syndrome, treated with 6 months of aliskiren vs. negative controls in patients with MFS under atenolol treatment. MRI for aortic pulsed wave velocity (PWV) and distensibility, measurements of central BP (CBP) and augmentation index (AIx) will be performed at the beginning and end of treatment. A blood drawn for serum markers of TGF-beta, extracellular matrix turnover and inflammation will also be performed at 0 and 6 months. We plan to determine whether aliskiren decreases aortic stiffness significantly more than negative controls in patients with MFS under atenolol treatment.

DETAILED DESCRIPTION:
Study design and study population The study design was a prospective randomized intervention study in a single center. A randomization process was performed to assign participants to either the aliskiren-treatment group or the negative control group in an open-label design. The duration of the study period was 24 weeks as the time frame for treatment. Duration of treatment was decided based on previous studies using RAS inhibitor 13,25. Aliskiren was administered to patients in the treatment group at an oral dose of 150-300 mg per day. Medication administration started after a baseline study with a dose of 150 mg of aliskiren, which was escalated to 300 mg of aliskiren at 4 weeks after evaluation of tolerability and the presence of adverse effects as angioedema, gastrointestinal symptoms, rash, gout, hypotension, and renal stones. The patients stopped taking aliskiren if serious adverse events such as angioedema or allergic reactions definitely related to the medication developed. Dose reduction was considered in cases with development of hyperkalemia, elevation of serum creatinine to twice baseline, symptomatic hypotension, gout, or renal stones. Dose reduction to 150 mg after escalation was performed on the decision of the investigators if the patient complained of discomfort and side effects that were probably related to the medication.

MFS patients were recruited at Samsung Medical Center from November 2009 to October 2014. All patients were receiving atenolol as standard β-blocker therapy. All patients gave written informed consent to participate in the study, which was approved by the Samsung Medical Center Ethics Committee. This trial is registered at ClinicalTrial.gov. (Identifier: NCT01715207) Inclusion criteria were age 14 to 55 years, a diagnosis of MFS by Ghent criteria, β-blocker treatment for at least 3 months, and no chronic RAS inhibitor therapy (i.e., angiotensin II receptor blockers or ACE inhibitors) for 90 days prior to screening. Exclusion criteria were previous medical history of aortic surgery and/or dissection, significant valve disease requiring surgery, aortic root dimension > 5.0 cm, renal dysfunction (creatinine > upper normal limit), pregnancy or planned pregnancy within 12 months of study entry or current breast feeding, known renal artery stenosis, hypersensitivity to aliskiren or any of the excipients, elevation of serum creatinine during follow-up (> 30% of baseline), diarrhea resulting in severe dehydration, development of gout or ureter stone, symptomatic hypotension (systolic blood pressure <90 mmHg with symptoms), hyperkalemia, and concomitant treatment with cyclosporin A.

Follow-up and outcomes All included patients were clinically followed to monitor adverse effects of angioedema, gastrointestinal symptoms, rash, gout, hypotension, and renal stone at initial examination, 1 week, 4 weeks, 8 weeks, 16 weeks, and 24 weeks. The following laboratory data were collected during the same period: potassium, electrocardiogram, creatinine, uric acid, and urine analysis. Echocardiographic evaluation, peripheral tonometric measurements of peripheral PWV, central aortic blood pressure and augmentation index, cardiac magnetic resonance imaging (cardiac MRI), and biomarkers were analyzed at baseline and after 24 weeks of treatment.

Safety information was collected, including all adverse events and all serious adverse events. Completion of a serious adverse event form was required for all serious adverse events that occurred during the study period. All serious adverse events were assessed by investigators and reported to the Novartis safety desk within 24 hours.

The primary end point was central aortic distensibility by cardiac MRI at 24 weeks, reported as the change over the 24-week period after randomization. The secondary end points were central aortic PWV by cardiac MRI, change in central aortic blood pressure (hereafter, aortic BP), augmentation index, peripheral PWV by tonometry, aortic root diameter by echocardiography, severity of aortic regurgitation by echocardiography, and dissection/rupture/operation of aneurysm.

Cardiovascular imaging - echocardiography and cardiac MRI Cardiac MRI Cardiac MRI was performed using a 1.5-Tesla scanner (Magnetom Avanto, Syngo MR; Siemens Medical Solutions, Erlangen, Germany). Aortic diameters were measured at four landmark levels: level 1, the ascending aorta at the level of bifurcation of the pulmonary artery; level 2, the upper descending thoracic aorta at the level of bifurcation of the pulmonary artery; level 3, the lower descending thoracic aorta at the level of the diaphragm; level 4, the abdominal aorta just above the iliac bifurcation. Cine imaging was also performed at the same levels to measure aortic stiffness.

Cardiac MRI analysis - central aortic distensibility and central aortic PWV Analyses of the MRIs were performed using commercial software (Argus version 4.02, Siemens Medical Systems, Germany) by experienced observers who were blinded to patient information. To measure central aortic distensibility, the systolic and diastolic cross-sectional areas were measured by manual contouring of the aorta through the cardiac cycle on the cine image. Distensibility at the four regions was calculated as the mean of values obtained from the following equation: Distensibility = (Amax - Amin)/[Amin × (Pmax - Pmin)](10-3mm/Hg), where Amax is the maximal (systolic) aortic area, Amin is the minimal (diastolic) aortic area, Pmax is the systolic blood pressure (SBP), and Pmin is the diastolic blood pressure (DBP). Central aortic blood pressure measured non-invasively by SphygmoCor was used for systolic and diastolic blood pressure.

Aortic PWV was measured according to the well-validated method using MRI 19. From the velocity-encoded MRIs, aortic contours were automatically detected and manually adjusted in each slice area throughout the cardiac cycle. The transit time between the flow curves of each region of the aorta was determined from the midpoint of the systolic up-slope on the flow versus time curve 26-28. The up-slopes were identified by drawing a line between the points of 40% and 60% maximum velocity on the waveform. The distance between each aortic level was measured on black blood images using a curved line along the center of the aorta. Based on these data, the regional PWV was calculated as the ratio of the distance between levels and the time differences between the arrival of the pulse wave at each level. The PWV was measured at two regions: the proximal aorta (proximal PWV between level 1 and level 2) and the entire aorta (PWV-total between level 1 and level 4).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MFS by Ghent criteria and/or genetically proven Fibrillin-1 (FBN1) mutation
2. Age between 14 and 55 years
3. Beta-blocker treatment at least 3 months
4. subjects must not have been receiving chronic RAS inhibitor therapy (i.e. ARBs, or ACE inhibitors)>= 90days prior to screening
5. Written informed consent from the patients or authorized representatives must be obtained

Exclusion Criteria:

1. previous medical history of aortic surgery and/or dissection
2. significant valve disease requiring surgery
3. aortic root dimension > 5.5 cm
4. renal dysfunction (creatinine > upper normal limit)
5. pregnancy or planned pregnancy within 12 months of study entry or breast feeding women
6. Known renal artery stenosis
7. Hypersensitivity to the aliskiren or to any of the excipients
8. Elevation of serum creatinine during follow-up (> 30% than baseline)
9. Diarrhea, resulting severe dehydration
10. Development of gout or ureter stone
11. Symptomatic hypotension (SBP<90 with symptom)
12. Hyperkalemia
13. Concomitant use with ciclosporin A

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Kyung Kim, PhD MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
to contact the principal investigator

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was premature termination due to the stop of supporting medication from company.
Groups:
- Atenolol & Aliskiren: Atenolol tablet and Aliskiren 150mg or 300mg tablet by mouth per day for 6month
  Aliskiren
  Atenolol
- Atenolol: Atenolol tablet(Negative controls, Open-label)
  Atenolol
Period: Overall Study
Arm/Group | Atenolol & Aliskiren | Atenolol
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atenolol & Aliskiren | Atenolol | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: yeaars] | 32.1 (9.3) | 33.2 (12.0) | 32.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Central Aortic Distensibility by MRI
Description: Analyses of the MRIs were performed using commercial software (Argus version 4.02, Siemens Medical Systems, Germany) by experienced observers who were blinded to patient information. To measure central aortic distensibility, the systolic and diastolic cross-sectional areas were measured by manual contouring of the aorta through the cardiac cycle on the cine image. Distensibility at the four regions was calculated as the mean of values obtained from the following equation: Distensibility = (Amax - Amin)/[Amin × (Pmax - Pmin)](10-3mm/Hg), where Amax is the maximal (systolic) aortic area, Amin is the minimal (diastolic) aortic area, Pmax is the systolic blood pressure (SBP), and Pmin is the diastolic blood pressure (DBP). Central aortic blood pressure measured non-invasively by SphygmoCor was used for systolic and diastolic blood pressure.
Time Frame: 6 months
Population: MFS patients were recruited at Samsung Medical Center from November 2009 to October 2014. All patients were receiving atenolol as standard β-blocker therapy.
Measure: Mean (Standard Deviation); unit: (mmHg ^ -1) x 10 ^ -3
Arm/Group | Atenolol & Aliskiren | Atenolol
Number analyzed (Participants) | 14 | 14
(mmHg ^ -1) x 10 ^ -3
  initial ascending aorta | 3.7 (1.3) | 4.7 (2.8)
  initial upper descending aorta | 5.7 (1.8) | 5.1 (2.5)
  initial lower descending aorta | 7.5 (2.7) | 6.3 (2.7)
  initial abdominal aorta | 2.4 (1.7) | 2.7 (1.3)
  follow up ascending aorta | 5.2 (2.7) | 5.0 (2.9)
  follow up upper descending aorta | 8.3 (4.7) | 6.0 (2.8)
  follow up lower descending aorta | 9.7 (4.6) | 7.1 (2.9)
  follow up abdominal aorta | 4.5 (3.4) | 3.5 (1.9)

2. Secondary Outcome: Central Aortic PWV(Pulsed Wave Velocity)
Description: Aortic PWV was measured according to the well-validated method using MRI 19. From the velocity-encoded MRIs, aortic contours were automatically detected and manually adjusted in each slice area throughout the cardiac cycle. The transit time between the flow curves of each region of the aorta was determined from the midpoint of the systolic up-slope on the flow versus time curve 26-28. The up-slopes were identified by drawing a line between the points of 40% and 60% maximum velocity on the waveform. The distance between each aortic level was measured on black blood images using a curved line along the center of the aorta. Based on these data, the regional PWV was calculated as the ratio of the distance between levels and the time differences between the arrival of the pulse wave at each level. The PWV was measured at two regions: the proximal aorta (proximal PWV between level 1 and level 2) and the entire aorta (PWV-total between level 1 and level 4).
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Atenolol and Aliskiren: Aliskiren (Norvatis) 300mg oral tablet
- Atenolol: Atenolol tablet(Negative controls, Open-label)
  Control group baseline 24 Weeks Central PWV (m/s)(26) by MRI regional PWV A (level 1-2) 3.8 (1.7) 3.6 (1.23) PWV-total (level 1-4) 5.0 (1.03) 4.9 (1.24)
Arm/Group | Atenolol and Aliskiren | Atenolol
Number analyzed (Participants) | 14 | 14
m/s
  baseline regional PWV A | 3.3 (1.03) | 3.8 (1.7)
  baseline PWV total | 4.5 (0.77) | 5.0 (1.03)
  follow up regional PWV A | 3.2 (0.8) | 3.6 (1.23)
  follow up PWV total | 4.7 (1.1) | 4.9 (1.24)

ADVERSE EVENTS:
Time Frame: 6months
Description: angioedema, GI symptom, rash, gout, hypotension, renal stone K, EKG, creatinine, uric acid, urine analysis Safety information will be collected including all AEs (adverse events) and all SAEs (Serious adverse events). Specially, a serious adverse event form should be completed for all serious adverse events during the study period. The serious adverse event will be checked by investigators. And investigators will report all SAEs to Novartis Safety desk within 24 hours since they know.
Groups:
- Atenolol & Aliskiren: Atenolol tablet and Aliskiren 150mg or 300mg tablet by mouth per day for 6month
  Treatment (n=14) Overall rate of adverse events 12 (85.7%) moderate to severe cases 0 generalized symptoms 8 (57.1%) gastrointestinal symptoms 4 (28.6%) lung problems 0 cardiovascular symptoms 3 (21.4%) central nervous system symptoms 5 (35.7%) Eye, nose, throat symptoms 4 (28.6%) gynecologic problems 1 (7.1%) problems of extremities 1 (7.1%)
- Atenolol: Atenolol tablet(Negative controls, Open-label)
  Control (n=14) Overall rate of adverse events 10 (71.4%) moderate to severe cases 2 (14.3%) generalized symptoms 4 (28.6%) gastrointestinal symptoms 3 (21.4%) lung problems 1 (7.1%) cardiovascular symptoms 0 central nervous system symptoms 1 (7.1%) Eye, nose, throat symptoms 1 (7.1%) gynecologic problems 1 (7.1%) problems of extremities 2 (14.3%)
Arm/Group | Atenolol & Aliskiren | Atenolol
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/14
Other Adverse Events (participants affected / at risk) | 8/14 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atenolol & Aliskiren (N=14) | Atenolol (N=14)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atenolol & Aliskiren (N=14) | Atenolol (N=14)
generalized symptoms (General disorders) | 8 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes